CLINICAL TRIAL: NCT06024733
Title: Effect of Total Intravenous Anesthesia by Targeted Controlled Infusion on Surgical Stress Response Compared to Inhalational Anesthesia
Brief Title: Intravenous Anesthesia by Targeted Controlled Infusion Versus Inhalational Anesthesia on the Surgical Stress Response
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Ali Galal, Assistant lecturer of Anesthesia, ICU and pain Relief South Egypt Cancer Institute- Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 525
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Total Intravenous Anesthesia; Inhalational Anesthesia; Surgical Stress Response; Target-controlled Infusion
MeSH Terms: interventions — Sevoflurane; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- inhalational (Sham Comparator)
  Interventions: Drug: Sevoflurane
- Target Controlled Infusion (Active Comparator)
  Interventions: Drug: Target Controlled Infusion
- Target Controlled Infusion and lidocaine (Active Comparator)
  Interventions: Drug: Target Controlled Infusion and lidocaine

INTERVENTIONS:
Drug: Sevoflurane — patient recieve propofol for induction and sevoflurane for maintenance
  Other Names: group 1
  Arms: inhalational
Drug: Target Controlled Infusion — target controlled infusion of propofol
  Other Names: GROUP 2
  Arms: Target Controlled Infusion
Drug: Target Controlled Infusion and lidocaine — patients will receive total intravenous anesthesia with propofol Target Controlled Infusion. At the induction of anesthesia, the patients will receive a bolus of lidocaine 1% 1.5 mg/kg and a continuous infusion of lidocaine 1% 2 mg/kg/h will be associated throughout the procedure.
  Other Names: GROUP3
  Arms: Target Controlled Infusion and lidocaine

SUMMARY:
This study aims to compare the effect of total Intravenous anesthesia Target-controlled infusion (TIVA-TCI) with inhalational anesthesia on stress response.

DETAILED DESCRIPTION:
Target-controlled infusion (TCI) techniques have been used to induce and maintain general anesthesia or to provide computer-assisted personalized sedation. Target-controlled infusion (TCI) systems are computer-assisted IV infusion pumps that use pharmacokinetic and pharmacodynamic mathematical modeling to maintain a user-designated target concentration at an effect site (typically the brain).

The clinician enters a desired target concentration for an anesthetic or another agent. The computer calculates the amount of the agent required to achieve the target concentration at the effect site and directs an infusion pump to deliver the calculated boluses or infusions. Therefore, TIVA-TCI allows a more stable hemodynamic profile during surgery, prevents long-acting opioid-induced accumulation and allows rapid recovery from general anesthesia.

Total intravenous anaesthesia (TIVA) regimen with Propofol is a useful anaesthetic technique, effectively controlling responses to tracheal intubation and intense surgical stimulation, while avoiding Inhalational anaesthetics and allowing rapid emergence from anaesthesia .

ELIGIBILITY:
Inclusion Criteria:

1. Patients subjected to lower abdominal cancer surgery.
2. Patients of both sexes
3. body mass index < 35 kg/m2.
4. Age from 18 to 60 years.
5. ASA, I-II.

Exclusion Criteria:

1. Patients with a history of severe cardiovascular or respiratory disease.
2. Severe hepatic, renal, or neurological diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The level of the stress response by serum level of insulin-like growth factors | Intraoperative and 24hours after surgery
  The serum level of insulin-like growth factors will be measured at preoperative, intraoperative after one hour of intubation, at the end of surgery and after extubation, and transfer to the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol, SAP
Time Frame: for one year after the end of study
Access Criteria: The data will be available upon a reasonable request from the corresponding author